CLINICAL TRIAL: NCT05601154
Title: Fluoride Bioavailability in Saliva After Use of Prescription and Over-the-counter Toothpastes Followed by Fluoride Mouthrinses
Brief Title: Fluoride in Saliva After Use of Fluoride Toothpastes Followed by Fluoride Mouthrinses
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Livia Tenuta, Associate Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: HUM00212598
Record Dates: First submitted 2022-10-26; First posted 2022-11-01 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — hydrated silica gel-based toothpaste

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Crest Cavity Protection (Active Comparator): Crest Cavity Protection toothpaste (1,100 ppm F) will be used to brush teeth, followed by a mouth rinse with tap water
  Interventions: Drug: Crest Cavity Protection toothpaste
- Crest Cavity Protection followed by Act Mint Fluoride Rinse (Active Comparator): Crest Cavity Protection toothpaste (1,100 ppm F) will be used to brush teeth, followed by a mouth rinse with Act Mint Fluoride Rinse (226 ppm)
  Interventions: Drug: Crest Cavity Protection toothpaste followed by Act Mint Fluoride Rinse
- Colgate PreviDent 5000+ (Active Comparator): Colgate PreviDent 5000+ (5,000 ppm F) will be used to brush teeth, followed by a mouth rinse with tap water
  Interventions: Drug: Colgate PreviDent 5000+ toothpaste
- Colgate PreviDent 5000+ followed by Act Mint Fluoride Rinse (Experimental): Colgate PreviDent 5000+ (5,000 ppm F) will be used to brush teeth, followed by a mouth rinse with Act Mint Fluoride Rinse (226 ppm)
  Interventions: Drug: Colgate PreviDent 5000+ toothpaste followed by Act Mint Fluoride Rinse

INTERVENTIONS:
Drug: Crest Cavity Protection toothpaste — Participants will brush their teeth with Crest Cavity Protection toothpaste (1,100 ppm F) for 1 minute, expectorate the foam, and rinse their mouths with 10 mL of tap water for 10 seconds
  Other Names: Over-the-counter fluoride toothpaste followed by water rinse
  Arms: Crest Cavity Protection
Drug: Crest Cavity Protection toothpaste followed by Act Mint Fluoride Rinse — Participants will brush their teeth with Crest Cavity Protection toothpaste (1,100 ppm F) for 1 minute, expectorate the foam, and rinse their mouths with 10 mL of Act Mint Fluoride Rinse (226 ppm) for 1 minute
  Other Names: Over-the-counter fluoride toothpaste followed by fluoride rinse
  Arms: Crest Cavity Protection followed by Act Mint Fluoride Rinse
Drug: Colgate PreviDent 5000+ toothpaste — Participants will brush their teeth with Colgate PreviDent 5000+ (5,000 ppm F) for 1 minute, expectorate the foam, and rinse their mouths with 10 mL of tap water for 10 seconds
  Other Names: Prescription fluoride toothpaste followed by water rinse
  Arms: Colgate PreviDent 5000+
Drug: Colgate PreviDent 5000+ toothpaste followed by Act Mint Fluoride Rinse — Participants will brush their teeth with Colgate PreviDent 5000+ (5,000 ppm F) for 1 minute, expectorate the foam, and rinse their mouths with 10 mL of Act Mint Fluoride Rinse (226 ppm) for 1 minute
  Other Names: Prescription fluoride toothpaste followed by fluoride rinse
  Arms: Colgate PreviDent 5000+ followed by Act Mint Fluoride Rinse

SUMMARY:
This study will evaluate fluoride (F) bioavailability in saliva when using an over-the-counter mouthrinse of 226 ppm F, immediately after brushing with an over-the-counter toothpaste of 1,100 ppm F or a prescription toothpaste of 5,000 ppm F. The study population will include twenty individuals, over the age of 18 years-old, from both genders, with normal oral health conditions and salivary flow rate, no need of urgent dental needs, from the Ann Arbor, MI area. Participants will be recruited from the University of Michigan School of Dentistry, in Ann Arbor, MI. Using a crossover design, twenty participants will be rotating through 4 different combinations of fluoride toothpaste (over-the-counter or prescription concentration) and fluoride mouth rinse (yes or no), in a 2 x 2 factorial design. Treatments to be tested will be as followed: Group #1 will brush with 1,100 ppm F (over-the-counter) toothpaste; Group #2 will brush with 1,100 ppm F (over-the-counter) toothpaste and rinse with over-the-counter 226 ppm F mouthrinse; Group #3 will brush with 5,000 ppm F (prescription) toothpaste; Group #4 will brush with 5,000 ppm F (prescription) toothpaste and rinse with over-the-counter 226 ppm F mouthrinse.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent form
* Participant understands and agrees to comply with the study protocol, and confirms availability for the entire duration of the study
* 18 years of age or older
* Good general health
* Good oral health, with no urgent treatment needs
* Normal salivary flow rate

Exclusion Criteria:

* Fail to understand or to agree to follow the study protocol
* Reduced salivary flow rate
* Poor general or oral health conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Area under the curve of fluoride bioavailability in saliva | 0 to 60 minutes after the interventions
  Fluoride concentration in saliva will be measured before (baseline) and up to 60 min after the interventions, and the area under the curve of fluoride concentration versus time will be calculated to estimate bioavailability

SECONDARY OUTCOMES:
Maximum fluoride concentration in saliva | 0 to 60 minutes after the interventions
  From the area under the curve, the time at which the concentration in saliva is highest will be determined

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dentistry, University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided